CLINICAL TRIAL: NCT03622567
Title: Assessing the Effect of Smartphone Push Notifications on Overall Score, Accuracy and Reaction Time of Brain Power Score
Brief Title: The Effect of Smartphone Push Notifications on Brain Power Score
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthTech Connex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HTC-BPS-001
Record Dates: First submitted 2018-08-01; First posted 2018-08-09 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Push Notifications (Other): Push notification number (0, 1, 3, 5) will be counter balanced within-subjects.
  Interventions: Behavioral: Smartphone push notifications

INTERVENTIONS:
Behavioral: Smartphone push notifications — The purpose of this study is to assess how smartphone push notifications can impact the overall score, accuracy and reaction time of participants using the Brain Power Score application (app). Push notification quantity will be varied and counter-balanced.

SUMMARY:
This study will examine how Brain Power Score, an objective measure of brain function, is affected by the presence of smartphone push notifications.

DETAILED DESCRIPTION:
Smartphones are a common device integrated into the lives of many individuals around the world. Researchers have previously found a relationship between mobile phone use and changes in brain activity, reaction times and sleep patterns.

Brain Power is a consumer-grade application using a proprietary combination of neurological (EEG) and behavioral (reaction time and accuracy) data to create a comprehensive score out of 1000 which allows users to have an objective evaluation of their brain performance.

This study will examine how Brain Power Score is affected by the presence of smartphone push notifications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* ≥19 years old
* Must be proficient in English
* Must be able to understand the study procedure and give informed consent

Exclusion Criteria:

* Unable to provide informed consent

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Total Brain Power Score | 20 minutes
  Brain Power Score combines neurological (EEG) and behavioral (reaction time and accuracy) data to create a comprehensive score out of 1000.

SECONDARY OUTCOMES:
Accuracy | 20 minutes
  Percentage of correctly classified instances
Reaction time | 20 minutes
  Time to respond to the stimulus (milliseconds)

CONTACTS AND LOCATIONS:
Locations (1):
- HealthTech Connex Centre for Neurology Studies, Surrey, British Columbia, Canada